CLINICAL TRIAL: NCT06248086
Title: A First-in-Human, Phase 1 Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of a Single-Induction Dose of convertibleCARTM-T Cells Armed With MicAbodyTM Protein (ASP2802) Followed by Maintenance Booster Doses of the MicAbody Protein in Patients With CD20-Positive Relapsed or Refractory B-Cell Lymphomas
Brief Title: A Study to Find a Suitable Dose of ASP2802 in People With CD20-positive B-cell Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The termination of the study was a business decision made by the sponsor.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2802-CL-0101
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: B-cell Lymphoma
Keywords: relapsed CD20-positive; refractory CD20-positive; CAR-T cell therapy; ASP2802
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: ASP2802 Low Dose followed by MA-20 (Experimental): Participants will receive a low dose of ASP2802 on Day 0 of cycle 1. Each participant will then receive up to 2 doses of MA-20 booster in each 28-day cycle.
  Interventions: Drug: ASP2802; Drug: MA-20
- Group B: ASP2802 Intermediate Dose followed by MA-20 (Experimental): Participants will receive an intermediate dose of ASP2802 on Day 0 of cycle 1. Each participant will then receive up to 2 doses of MA-20 booster in each 28-day cycle, with dose level(s) selected from Group A.
  Interventions: Drug: ASP2802; Drug: MA-20
- Group C: ASP2802 High Dose followed by MA-20 (Experimental): Participants will receive a higher dose of ASP2802 on Day 0 of cycle 1. Each participant will then receive up to 2 doses of MA-20 booster in each 28-day cycle, with dose level(s) selected from Group B.
  Interventions: Drug: ASP2802; Drug: MA-20

INTERVENTIONS:
Drug: ASP2802 — Intravenous (IV) infusion
  Other Names: MACT
Drug: MA-20 — IV infusion
  Other Names: ASP101G; MicAbody

SUMMARY:
CAR-T cell therapy is a type of treatment for people with certain lymphomas. T-cells are white blood cells that help to fight infections. CAR-T cell therapy improves the body's T-cells to help them better fight cancer cells.

ASP2802 is a type of CAR-T cell therapy given with MA-20. MA-20 is a protein that helps the CAR-T cell therapy work inside the body.

Before ASP2802 is available as a treatment, the researchers need to understand how it is processed by and acts upon the body. This information will help find a suitable dose for future studies and check for potential medical problems from the treatment.

In this study, ASP2802 is being tested in humans for the first time. ASP2802 has already been tested in the laboratory and in animals. This is the standard way new potential treatments are developed.

People taking part in this study will be adults with CD20-positive B-cell lymphomas. CD20 is a protein found on a type of white blood cell called a B-cell. Some people with B-cell lymphomas have more CD20 on these cells. Their cancer will have come back after it had disappeared with earlier therapy (relapsed) or it will have become resistant to previous treatment (refractory).

The main aims of the study are to check the safety of ASP2802, how well it is tolerated, and to find a suitable dose of ASP2802.

This is an open-label, adaptive study. Open-label means that people in this study and clinic staff will know that people will receive ASP2802 treatment. Adaptive means the treatments may change, depending on earlier results in the study.

There will be 3 groups of people in this study and 3 doses of ASP2802. Groups A, B and C will receive ASP2802 treatment. Group A will start treatment first with a low dose of ASP2802. If Group A tolerates the low dose of ASP2802, then Group B will receive the higher dose of ASP2802. If Group B tolerates the higher dose of ASP2802, then Group C will receive the highest dose of ASP2802.

There are several steps in this treatment. First, T-cells are removed from the blood by inserting a small tube (cannula) into a vein and connecting it to a machine that separates out the blood cells. The machine collects the T-cells and returns the rest of the blood cells back into the bloodstream. The collected T-cells are sent to the lab to be changed into improved T-cells (with ASP2802) to fight the cancer. This may take several weeks, so people in the study may receive extra treatment, to keep the cancer under control during this time.

Before the improved T-cells go back in the body, people will visit the clinic so that the study doctors can do a series of checks to make sure they are well enough to receive the T-cells. A few days before the improved T-cells go back into the body, people in the study will have chemotherapy for 3 days. This is to make sure the cancer is at its lowest level before people are treated with ASP2802. Then, the improved T-cells are fed back into the bloodstream using a drip attached to the cannula. After this, a booster of MA-20 will be given at the set dose by infusion on Day 3 and Day 17 in a 28-day cycle. If people respond well to treatment, they may stay on the same dose during the next cycle; if they have medical problems from the treatment, they may get a lower dose during the next cycle. The next group of people may receive a different dose (higher or lower) of MA-20 depending on the results from the previous group. People in the study will continue receiving MA-20 in this way until: they have certain medical problems from the treatment on the lowest dose of MA-20; they start other cancer treatment; their cancer gets worse; they or the study doctor decides they should stop treatment; they do not come back for treatment.

After treatment has finished, people in the study will visit the clinic regularly for 2 years and continue to be monitored for up to 15 years.

Some people may be treated again with MA-20. This may happen for people who have responded to treatment and then relapse within a year, or for people that have a partial response and have a slow growing lymphoma.

During the study, people will visit the study hospital many times. During most visits, the study doctors will do a medical examination, blood tests and check vital signs. Vital signs include temperature, breathing rate, blood pressure, blood oxygen levels, and heart rate. They will also check for medical problems. In some visits, computerized tomography (CT) scans and electrocardiograms (ECGs) to check the heart rhythm will also be done.

People will have several hospital stays during their treatment. This may be during their chemotherapy, then from Days -1 to 7 and Days 17 to 21 during the cycle 1 of MA-20. Day -1 means 1 day before treatment with ASP2802. During this time, people will be closely monitored for medical problems, have EGCs and have a biopsy taken. During the extra cycles of MA-20, there will be the option of staying overnight.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically-confirmed cluster of differentiation (CD) 20-positive B-cell lymphoma (CD20 expression should be demonstrated by local testing at the time of relapse or progression and within 1 month of study screening) which may include the following aggressive large cell or indolent subtypes.

  * Diffuse large B-cell lymphoma (DLBCL), Not otherwise specified (NOS)
  * Follicular lymphoma grade 3B
  * Primary mediastinal large B-cell lymphoma
  * T-cell/histiocyte-rich large B-cell lymphoma
  * DLBCL associated with chronic inflammation
  * Intravascular large B-cell lymphoma
  * Anaplastic lymphoma kinase fusion gene (ALK)+ large B-cell lymphoma
  * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma
  * High grade B-cell lymphoma with proto-oncogene located on chromosome 8 (MYC) and B-cell leukemia/lymphoma 2 gene (BCL2) and/or B-cell leukemia/lymphoma 6 gene (BCL6) rearrangements
  * High-grade B-cell lymphoma, NOS
  * Human herpes virus type 8 (HHV8)+ DLBCL, NOS
  * Primary cutaneous DLBCL, leg type
  * Transformed follicular lymphoma
  * Follicular lymphoma
  * Marginal zone lymphoma
* Participant has either relapsed or refractory disease defined as:

  * Relapse after ≥ 2 prior lines of therapy; or
  * Refractory disease: After ≥ 2 prior lines of therapy and did not achieve complete response (CR)
* Participants who have undergone autologous stem cell transplant (SCT) with disease progression or relapse following SCT will be eligible if all other eligibility criteria are met.
* Participants with lymphoma must have evaluable or measurable disease according to the Lugano criteria for response assessment of lymphoma. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
* At least 2 weeks or 5 half-lives, whichever is longer, must have elapsed since any prior anticancer therapy at the time of leukapheresis, except for inhibitory/stimulatory immune checkpoint therapy, which requires 3 half-lives.

Exceptions:

* There is no time restriction with regard to prior intrathecal chemotherapy (including steroids) provided there is complete recovery from any acute toxic effects of such.
* Participants receiving steroid therapy at physiologic replacement doses (≤ 5 milligrams per day (mg/day) of prednisone or equivalent doses of other corticosteroids) are allowed. Use of higher doses of systemic steroids must stop at least 72 hours before leukapheresis.
* Radiation therapy must have been completed at least 2 weeks prior to leukapheresis.

  * Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities, such as alopecia, nutritional support measures, electrolyte abnormalities or those not impacting the investigator's ability to assess treatment-emergent toxicities).
  * Participant has cardiac ejection fraction (EF) ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an echocardiogram or multigated acquisition scan (MUGA) and no clinically significant ECG findings.
  * Participant has no clinically significant pleural effusion.
  * Participant has baseline oxygen saturation > 90% on room air at rest.
  * Participant has a life expectancy of ≥ 12 weeks.
  * Participant has an ECOG performance score of 0, 1 or 2.
  * Female participant is not pregnant and at least 1 of the following conditions apply:
* Not a woman of childbearing potential (WOCBP).
* WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 6 months after final study treatment administration.

  * Female participant must agree not to breastfeed starting at screening and throughout the study period and for 6 months after final study treatment administration.
  * Female participant must not donate ova starting at first dose of IP and throughout the study period and for 6 months after final study treatment administration.
  * Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 6 months after final study treatment administration.
  * Male participant must not donate sperm during the treatment period and for 6 months after final study treatment administration.
  * Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 6 months after final study treatment administration.
  * Participant agrees not to participate in another interventional study while participating in the present study
  * Participant has adequate organ function at baseline. If a participant has received a recent blood transfusion, the laboratory tests must be obtained ≥ 28 days after any blood transfusion.

Additional Inclusion Criteria prior to Lymphodepletion Chemotherapy:

* Participant has adequate hepatic function defined by aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); total bilirubin ≤ 1.5 × ULN (participants with Gilbert's syndrome may be included if their total bilirubin is ≤ 3.0 × ULN and direct bilirubin is ≤ 1.5 × ULN)
* Participant has adequate renal function defined by:

  * Creatinine < 1.5 × ULN, or
  * An estimated creatinine clearance (CrCl) of ≥ 60 milliliter per minute (ml/min) as calculated by the Cockcroft-Gault equation
* Participant has adequate bone marrow function defined by absolute neutrophil count ≥ 500/microliter (µl) and platelet count ≥ 50 000/µl (unless inadequate bone marrow function is thought to be related to bone marrow involvement with the lymphoproliferative neoplasm).

Exclusion Criteria:

* Participant has been diagnosed with the following conditions:

  * B-lymphoblastic leukemia/lymphoma (B-ALL/LBL)
  * chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL)
  * Burkitt lymphoma
  * Richter's transformation of CLL/SLL
  * Epstein-Barr virus (EBV)+ DLBCL, NOS
  * Mantle cell lymphoma
* Known history or suspicion of central nervous system involvement by lymphoma.
* Participant weighs < 45 kilograms (kg) at screening.
* Participant had prior allogeneic hematopoietic stem cell transplantation (HSCT).
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has a history of non-study related malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast) unless disease free for at least 3 years.
* Participant has a history of myocardial infarction, cardiac angioplasty or stenting, unstable angina or other clinically significant cardiac disease within 12 months of enrollment or has cardiac atrial or cardiac ventricular lymphoma involvement.
* Participant has known abnormal lung function: forced expiratory volume (FEV) < 60% prediction, diffusing capacity of the lung for carbon monoxide < 60% prediction, blood oxygen saturation < 90% on room air.
* Participant has intracranial hypertension or unconsciousness, respiratory failure or disseminated intravascular coagulation.
* Participant has leukocytosis (white blood cell [WBC] count ≥ 25 000/µL) or rapidly progressive disease that would compromise ability to complete study therapy.
* Participant has a history or presence of a central nervous system (CNS) disorder such as cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, seizure disorder or autoimmune disease with CNS involvement that may impair the ability to evaluate neurotoxicity.
* Participant has any of the following per screening serology test:

  * Hepatitis A virus (HAV) antibodies immunoglobulin M (IgM)
  * Positive hepatitis B surface antigen (HBsAg) or detectable hepatitis B Deoxyribonucleic acid (DNA). Participants with negative HBsAg, positive hepatitis B core antibody (anti-HBc) and negative anti-HBs are eligible if hepatitis B DNA is undetectable
  * hepatitis C virus (HCV) antibodies unless HCV ribonucleic acid (RNA) is undetectable
* Participant has human immunodeficiency virus (HIV) per screening serology test.
* Participant has a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) polymerase chain reaction (PCR) test at Screening.
* Participant has a primary immunodeficiency or history of systemic autoimmune disease (e.g., Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/disease-modifying agents within the last 2 years.
* Participant has presence of fungal, bacterial (e.g., tuberculosis), viral or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple infections like urinary tract infections and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
* Participant's adverse reactions (excluding alopecia or vitiligo) from prior therapy have not improved to Grade 1 or baseline at least 14 days prior to Screening.
* Participant has received rituximab within 14 days prior to Screening.
* Participant has presence of any other concurrent medical condition or factors that would prevent the participant from undergoing or completing protocol-specified treatment, or makes the participant unsuitable for study participation.
* Participant had prior treatment with CD20 CAR-T cell or CD20 bi-specific therapy.
* Participant has a known or suspected hypersensitivity to ASP2802 (MACT), MA-20, fludarabine, cyclophosphamide or any components of the formulations used.
* Participant is receiving treatment with anticoagulants.

Additional Exclusion Criteria required for Lymphodepletion Chemotherapy:

* Participant received bridging therapy within 10 days prior to start of lymphodepletion chemotherapy (LDC).
* Participant has an active systemic infection present or onset of fever ≥ 38°C/100.4°F, not related to underlying disease. Participants who meet either of these on the day of scheduled ASP2802 (MACT) infusion should have ASP2802 (MACT) administration delayed.
* Participant has a positive SARS-CoV-2 PCR test.
* Participant has an intercurrent illness or toxicity that would place the participant at undue risk of proceeding to LDC and ASP2802 (MACT) infusion.
* Participant is receiving therapeutic doses of corticosteroids (defined as ≥ 20 mg/day prednisone or equivalent) within 24 hours prior to LDC. Physiologic replacement, topical, intranasal and inhaled steroids are permitted.
* Participant has signs of pre-existing CNS disease or toxicity.
* Participant has had major surgery within 28 days prior to the start of study treatment.
* Participants should not experience a significant worsening in clinical status compared to initial eligibility criteria that would increase the risk of adverse events associated with LDC or ASP2802 (MACT) infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 10 months
  A DLT is defined as any event meeting the DLT criteria occurring within 28 days after ASP2802 (MACT) infusion and/or 28 days after the first dose of each administered dose of MA-20 during the dose escalation phase not attributable to a cause other than investigational product (IP).
Number of participants with Adverse Events (AEs) | Up to 26 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study IP, whether or not considered related to the study IP and other study treatments.
  Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study IP and other study treatments. This includes events related to the (study) procedures.
Number of participants with Serious Adverse Events (SAEs) | Up to 26 months
  A Serious Adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other medically important event.
Number of participants with laboratory value abnormalities and/or AEs | Up to 26 months
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with vital sign abnormalities and/or AEs | Up to 26 months
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 26 months
  Number of participants with potentially clinically significant ECG values.
Number of Participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status scores | Up to 26 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP2802 in blood: Maximum Concentration (Cmax) | Up to 26 months
  Cmax will be recorded from the PK blood samples collected.
PK of ASP2802 in blood: Time to maximum concentration (tmax) | Up to 26 months
  tmax will be recorded from the PK blood samples collected.
PK of ASP2802 in blood: Area under the concentration-time curve (AUC)0-28d | Up to 26 months
  AUC0-28d will be recorded from the PK blood samples collected.
PK of ASP2802 in blood: concentration | Up to 26 months
  Concentration will be recorded from the PK plasma samples collected.
PK of MA-20 in serum: Cmax | Up to 26 months
  Cmax will be recorded from the PK serum samples collected.
PK of MA-20 in serum: tmax | Up to 26 months
  tmax will be recorded from the PK serum samples collected.
PK of MA-20 in serum: Trough concentration (Ctrough) | Up to 26 months
  Ctrough will be recorded from the PK serum samples collected.
PK of MA-20 in serum: AUC0-14d | Up to 26 months
  AUC0-14d will be recorded from the PK serum samples collected.
PK of MA-20 in serum: Apparent terminal half-life (t1/2) | Up to 26 months
  t1/2 will be recorded from the PK serum samples collected.
PK of MA-20 in serum: Apparent terminal elimination rate constant (Kel) | Up to 26 months
  Kel will be recorded from the PK serum samples collected.
PK of MA-20 in serum: Clearance (CL) | Up to 26 months
  CL will be recorded from the PK serum samples collected.
Number of participants with positive anti-drug antibodies to MA-20 | Up to 26 months
Objective Response Rate (ORR) of ASP2802 per Lugano Response Criteria | Up to 26 months
  ORR is defined as the proportion of participants whose best overall response is a Complete Response (CR) or Partial Response (PR).
Best Overall Response (BOR) of ASP2802 per Lugano Response Criteria | Up to 26 months
  BOR is defined as the proportion of participants achieving CR or PR based on the Lugano Treatment Response Criteria for NHL.
Duration of Response (DOR) of ASP2802 per Lugano Response Criteria | Up to 26 months
  DOR is defined as the time from the date of first documented response (CR or PR) to the date of first documented disease progression (PD) or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) of ASP2802 | Up to 26 months
  PFS is defined as time from start of treatment to progressive disease (PD) or death from any cause, whichever occurs first.
Overall Survival (OS) of ASP2802 | Up to 88 months
  OS is defined as is defined as time from start of ASP2802 to death.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Site AU61004, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.